CLINICAL TRIAL: NCT07043933
Title: The Effect of a Mobile-Compatible Web-Based Hydration Tracking Program on Hydration Knowledge, Attitudes, and Behaviors in Older Adults: A Randomized Controlled Trial
Brief Title: Effect of a Mobile-Based Hydration Tracking Program on Knowledge, Attitudes, and Behaviors in Older Adults
Acronym: SIVI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ezgi Atasoy (Other)
Responsible Party: Sponsor-Investigator, Ezgi Atasoy, Lecturer (Part-Time), Dokuz Eylul University
Organization: Dokuz Eylul University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: DEU-HYDRO-RCT-2025-01
Record Dates: First submitted 2025-06-21; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Dehydration; Older Adults (65 Years and Older); Hydration Status; Self-management Behavior; Mobile Application; Web Based Intervention
Keywords: Dehydration; Aged; Hydration; Older Adults; Mobile Applications; Self-Management
MeSH Terms: conditions — Dehydration

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either the intervention group, which receives the mobile-compatible web-based hydration application, or the control group, which receives standard education. Each group will be followed in parallel for 8 weeks.
Who Masked: Outcomes Assessor
Masking Description: Only the outcomes assessor (data analyst/statistician) is blinded to the allocation of participants to reduce the risk of bias.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Intervention Group (Experimental): Participants in this group will receive individualized face-to-face training and use the mobile-compatible, web-based hydration tracking application (SIVI) daily for 8 weeks. They will receive reminders, set personalized fluid intake goals, track their daily intake using visual tools, and access educational materials through the app. A standard water bottle will also be provided for consistent measurement.
  Interventions: Behavioral: Mobile-Compatible Web-Based Hydration Tracking Program
- Arm 2: Control Group (No Intervention): Participants in this group will receive rutine care. They will not receive access to the SIVI application or any structured follow-up. A standard water bottle will also be provided for intake tracking purposes.

INTERVENTIONS:
Behavioral: Mobile-Compatible Web-Based Hydration Tracking Program — Intervention Description:
  The SIVI Hydration Application is a mobile-compatible, web-based behavioral intervention designed specifically for older adults. It supports self-monitoring and self-management of daily fluid intake through features such as personalized fluid goals, visual drink-logging with icons, daily reminders, progress graphics, educational videos, and motivational digital badges. The app was developed using gerotechnology and universal design principles to accommodate cognitive and sensory changes common in aging. Its unique focus on hydration behavior, combined with usability features like large fonts, high contrast, and voice-assisted guidance, distinguishes it from general health or diet tracking apps. Participants use the app for 8 weeks as part of a structured intervention with training and weekly follow-up.
  Other Names: SIVI Mobile Hydration Tracker; SIVI Hydration Application
  Arms: Arm 1: Intervention Group

SUMMARY:
This randomized controlled trial aims to evaluate the impact of a mobile-friendly, web-based hydration tracking application (named "SIVI") on hydration-related knowledge, attitudes, and behaviors in older adults. Inadequate fluid intake is a common and modifiable risk factor for dehydration in the elderly, leading to increased morbidity, hospitalizations, and functional decline. However, many older individuals forget to drink fluids or face barriers such as fear of incontinence, mobility limitations, or cognitive challenges.

This study will include 70 community-dwelling older adults aged 65-84 years, recruited from a Family Health Center. Participants will be randomly assigned to either the intervention or control group. The intervention group will use the SIVI application for two months. The app is specially designed for older adults and includes features such as personalized fluid goals, reminders, hydration education modules, feedback, and a user-friendly interface with large fonts and high contrast. Participants will log their daily fluid intake, receive motivational messages, and access videos and information about healthy hydration habits. A water bottle will be provided to standardize measurement across groups.

The control group will receive only routine care. Both groups will complete questionnaires measuring demographics, hydration knowledge, attitudes, behaviors, and fluid consumption habits at baseline, one month, and two months.

Data collection will be conducted face-to-face by the researcher, and analysis will be performed using SPSS 22.0. Statistical tests will include descriptive statistics, Shapiro-Wilk for normality, chi-square for categorical data, and t-tests and ANOVA for comparisons over time.

The results are expected to show that the SIVI application improves older adults' hydration knowledge, fosters positive attitudes, and promotes healthy fluid intake behaviors, thus supporting self-management of hydration and potentially reducing dehydration-related health risks.

DETAILED DESCRIPTION:
1.1 Definition and Importance of the Problem Maintaining adequate fluid intake is a critical component of health across all stages of life. Proper hydration is essential for regulating blood pressure, enabling biochemical reactions, supporting nutrient digestion and absorption, maintaining cell and tissue function, thermoregulation, joint lubrication, and the elimination of toxins from the body (Armstrong & Johnson, 2018; Lorenzo et al., 2019; Li et al., 2023).

In older adults, various physiological and behavioral changes make it difficult to maintain adequate hydration. These include a diminished sense of thirst, reduced total body water, forgetfulness, aversion to the taste of water, fear of incontinence, and difficulty accessing fluids due to mobility issues. Such factors often lead to insufficient hydration and, eventually, to dehydration (Masot et al., 2020; Mentes & Gaspar, 2020; Dmitrieva et al., 2024).

Dehydration is a common condition among the older adults, particularly in institutional settings, and is associated with numerous negative health outcomes. These include headaches, dizziness, urinary tract infections, constipation, medication toxicity, respiratory infections, reduced muscle strength, delayed wound healing, fatigue, increased risk of falls, and cognitive impairment (Paulis et al., 2022; Parkinson et al., 2023; Purvis & Gion, 2024). In addition to increasing morbidity and mortality, dehydration extends hospital stays and increases readmission rates (Edmonds et al., 2021; Beck et al., 2021).

In Türkiye, studies indicate that approximately one in three individuals over the age of 65 attending outpatient clinics show signs of dehydration. Factors such as female gender, low education level, diabetes mellitus, and chronic kidney disease have been found to be associated with higher dehydration risk. Dehydrated individuals are also more likely to experience reduced physical functioning, sarcopenia, and falls (Atcıyurt et al., 2023).

While dehydration is often preventable, older adults may face challenges in recognizing or responding to their hydration needs. However, consistent daily fluid intake and regular monitoring can significantly reduce the risk. Hence, effective hydration self-management strategies are crucial for maintaining health and preventing complications among older adults (Jimoh et al., 2015; Garcia, 2022; Syed et al., 2024).

Recent interventions based on self-monitoring and digital support, such as wearable devices and mobile apps, have shown promising results. While there are some Turkish studies evaluating the effectiveness of education and auditory reminders (e.g., smartwatches) in nursing home residents (Çetin & Eşer, 2022), there is a lack of randomized trials focused on mobile health apps specifically tailored for older adult users in Türkiye.

Mobile health (mHealth) applications can support older adults by helping them monitor their fluid intake independently and consistently. Compared to smartwatches, mobile apps offer broader interactivity, greater visual clarity, and more accessible learning tools including videos, infographics, and personalized feedback (Siette et al., 2020). Apps also provide reminders and motivational tools that can promote sustained behavioral change.

In this context, the mobile-compatible, web-based hydration tracking application "SIVI" was developed to help older adults monitor their fluid intake, learn about hydration, and receive personalized feedback. Designed using principles of gerotechnology and age-friendly usability, SIVI features large fonts, high-contrast colors, customizable daily fluid targets, visual feedback tools, educational videos, and a question-and-answer interface with the researcher.

SIVI's usability and design were informed by prior literature, expert input, and pilot testing with older adults. The program aims to empower older adults to take a more active role in managing their hydration, thereby improving health outcomes and quality of life.

1.2 Aim of the Study This study aims to examine the effect of a mobile-compatible, web-based hydration tracking program developed for older adults on their hydration knowledge, attitudes, behaviors, and daily fluid intake.

1.3 Research Question and Hypotheses Research Question: Does the use of the mobile-compatible, web-based hydration tracking application (SIVI) improve daily fluid intake and hydration-related knowledge, attitudes, and behaviors among older adults? Null Hypothesis (H0): There is no statistically significant difference between the intervention and control groups in hydration knowledge, attitude, behavior, and fluid intake scores after the intervention.

Alternative Hypotheses:

• H1: There will be a statistically significant increase in hydration knowledge scores in the intervention group compared to the control group.

• H2: There will be a statistically significant increase in hydration attitude scores in the intervention group compared to the control group.

* H3: There will be a statistically significant increase in hydration behavior scores in the intervention group compared to the control group.
* H4: There will be a statistically significant increase in daily fluid intake in the intervention group compared to the control group.

  2. MATERIALS AND METHODS 2.1 Study Design This study is designed as a single-blind, block-randomized controlled trial. The aim is to assess the impact of the SIVI mobile-compatible web-based hydration tracking program on hydration knowledge, attitudes, behaviors, and fluid intake among community-dwelling older adults. The study will be conducted between October 2025 and March 2026 at Mehmet Fevzi Özsaruhan No. 24 Family Health Center in İzmir, Türkiye. Participants will be randomly assigned to either the intervention or control group in equal numbers using block randomization. To prevent bias, the statistician conducting data analysis will be blinded to group allocation.

2.2 Population and Sampling The study population will include individuals aged 65 to 84 years who live in the community and meet the inclusion criteria. A power analysis indicated that a sample of 26 individuals per group (total n=52) would provide 80% power to detect a moderate effect size. To account for potential dropouts, the sample size was increased to 35 participants per group (total n=70).

Inclusion Criteria:

• Aged 65 to 84 years

* Primary school education or higher
* Cognitive, sensory, and motor abilities sufficient for mobile phone use
* Willing to participate in the study
* Owns a mobile phone compatible with the application
* Daily fluid intake below ESPEN guidelines (≤2.0 L/day for men, ≤1.6 L/day for women)

Exclusion Criteria:

* Diagnosed with urinary incontinence
* Neurological or psychiatric disorders affecting mental status
* Severe hearing, vision, or speech impairments
* Diagnosed illnesses affecting fluid intake (e.g., kidney failure, heart failure)
* Swallowing difficulties
* Limited ability to perform basic activities of daily living
* Interruption in app use for one week or more
* Health conditions that may affect hydration needs during follow-up 2.3 Data Collection Tools

The following validated and researcher-developed instruments will be used for data collection:

* Descriptive Characteristics Form
* Fluid Intake Habits Form
* Hydration Knowledge, Attitudes, and Behaviors Scale (HyKS): Adapted to Turkish through a rigorous translation-back translation process with expert review (Veilleux et al., 2020).
* System Usability Scale (SUS): Administered to the intervention group only at the end of the study 2.4 Intervention: SIVI Application

The intervention group will receive face-to-face training and install the SIVI app, which they will use for eight weeks. Features of the app include:

* Personalized fluid intake targets
* Daily reminders
* Visual intake diary with cup/bottle icons
* Progress tracking graphics
* Educational videos and text modules
* A secure Q&A platform with the researcher
* Feedback via digital badges when daily goals are met Participants in both groups will receive the same model of water bottle to facilitate standardized self-monitoring. Weekly follow-up calls and twice-daily SMS reminders will be used to reinforce app use in the intervention group. A family physician will monitor participants' health status throughout the intervention to ensure safety.

The control group will receive only routine care services. They will not use the app.

2.5 Data Collection Procedure

Data will be collected at three points:

• Baseline (Day 0): Informed consent, demographic data, HyKS, Fluid Intake Habits Form

* Midpoint (1 Month): Repeat HyKS and habits form, app usage data automatically extracted
* Post-test (2 Months): Final data collection, including SUS for the intervention group Daily app usage is expected to take less than five minutes. 2.6 Data Analysis Statistical analysis will be performed using SPSS version 22.0. The Shapiro-Wilk test will assess normality. Depending on distribution characteristics, Student's t-tests or Mann-Whitney U tests will be used for between-group comparisons. Repeated measures ANOVA or Friedman tests will analyze within-group changes over time. Chi-square tests will be applied for categorical variables. Significance will be set at p<0.05.

  3. ETHICAL CONSIDERATIONS AND LIMITATIONS 3.1 Ethical Considerations This study was approved by the Non-Interventional Research Ethics Committee. All procedures will be conducted in accordance with the Declaration of Helsinki and relevant national regulations. Written informed consent will be obtained from all participants prior to inclusion in the study.

Participation in the study is entirely voluntary, and participants are free to withdraw at any time without any consequences. Confidentiality and anonymity of the data will be strictly maintained. The application's backend will store data on encrypted servers compliant with Personal Data Protection Law.

The study does not involve any invasive procedures, and there are no known significant physical risks associated with participation. Participants can mute reminders or exit the app at any time.

A family physician on the research team will monitor participants for adverse events such as vomiting, fever, or upper respiratory tract infections. If any clinical condition arises that could affect hydration needs, the physician will advise whether the participant should pause app use.

3.2 Limitations Several limitations must be acknowledged in interpreting the study findings. First, the study is single-center and conducted only in İzmir, Türkiye, which may limit the generalizability of results to other regions or populations. Second, the sample is restricted to individuals who own smartphones and are digitally literate. Third, the follow-up period is limited to two months, and long-term effects of the intervention will not be evaluated.

Additionally, standardized bottles and visual diary features in the intervention group aim to minimize measurement variability. Lastly, outcome assessors and the data analyst will remain blinded to reduce risk of bias.

4. CONTRIBUTIONS 4. Scientific and Practical Contributions

This study is expected to make several contributions to the field of geriatric health and mobile health (mHealth) interventions:

1. Innovation in Geriatric Care: This is the first randomized controlled trial in Türkiye to evaluate the effects of a mobile-compatible web-based hydration tracking program specifically developed for older adults. It offers a novel approach to behavioral change in hydration through digital self-management.
2. Contribution to Evidence-Based Practice: The findings of this study will contribute to the growing body of evidence supporting the use of mobile health technologies for promoting healthy behaviors in aging populations. If effective, the intervention may be integrated into routine primary care and geriatric services.
3. Public Health Impact: Improved hydration behaviors can lead to reduced risk of preventable health complications such as urinary tract infections, falls, and hospitalizations, thereby enhancing older adults' quality of life and reducing healthcare costs.
4. Usability Insights: The study will provide insights into the usability and acceptability of digital health tools among older adults in Türkiye, helping guide future development of age-friendly mobile applications.
5. Scalability and Dissemination: The modular structure of the SIVI application and its web-based delivery model support easy scalability and adaptation to different regions and languages, making it suitable for use in diverse older adults.

5. CONCLUSION This study addresses an urgent and under-recognized public health issue-dehydration among older adults-through the development and testing of a mobile-compatible, web-based hydration tracking application named SIVI. Given the high prevalence of dehydration in this population and its association with multiple adverse health outcomes, innovative solutions that promote hydration self-management are needed. The SIVI application, designed with age-appropriate features and content, represents a practical, scalable, and evidence-informed approach to digital health promotion By combining behavioral theory, gerontological principles, and user-centered technology design, the intervention aims to foster meaningful changes in hydration knowledge, attitudes, and daily habits. If successful, the program will support community-dwelling older adults in meeting their daily fluid intake needs, potentially preventing complications and enhancing overall well-being.

The study's design-a single-blind, block-randomized controlled trial-ensures methodological rigor and enhances the validity of its findings. The use of validated measurement tools, real-time tracking, and usability assessments strengthens the study's reliability. Moreover, ethical principles and participant safety are prioritized throughout the intervention period, supported by routine health monitoring by a qualified physician The findings from this research are expected to make a significant contribution to the fields of geriatric nursing, health informatics, and public health. The results could inform future interventions, contribute to policy development on older care and digital inclusion, and inspire further innovation in mobile health tools designed for vulnerable populations Ultimately, this study demonstrates how digital tools, when thoughtfully designed and evidence-based-can empower older adults to take control of their health in simple but impactful ways.

6.REFERANCES

1. Atasoy, E., Akyol, M. A., Söylemez, B. A., & Küçükgüçlü, Ö. (2025). Effectiveness of Self-Hydration Management Interventions in Middle-Aged and Older Adults: A Systematic Review and Meta-Analysis. Journal of gerontological nursing, 51(5), 17-25. https://doi.org/10.3928/00989134-20250326-01
2. Armstrong, L. E., & Johnson, E. C. (2018). Water Intake, Water Balance, and the Elusive Daily Water Requirement. Nutrients, 10(12), 1928. https://doi.org/10.3390/nu10121928
3. Atciyurt, K., Heybeli, C., Smith, L., Veronese, N., & Soysal, P. (2024). The prevalence, risk factors and clinical implications of dehydration in older patients: a cross-sectional study. Acta clinica Belgica, 79(1), 12-18. https://doi.org/10.1080/17843286.2023.2275922 3. Beck, A. M., Seemer, J., Knudsen, A. W., & Munk, T. (2021). Narrative Review of Low- Intake Dehydration in Older Adults. Nutrients, 13(9), 3142. https://doi.org/10.3390/nu13093142
4. Cetin, P., & Eser, I. (2022). Effect of an Audible Alarm on the Fluid Consumption of Older Adults Living in a Nursing Home: A Randomized Controlled Trial. Journal of gerontological nursing, 48(9), 39-46. https://doi.org/10.3928/00989134-20220808-02
5. Dmitrieva, N. I., Boehm, M., Yancey, P. H., & Enhörning, S. (2024). Long-term health outcomes associated with hydration status. Nature reviews. Nephrology, 20(5), 275-294. https://doi.org/10.1038/s41581-024-00817-1
6. Edmonds, C. J., Foglia, E., Booth, P., Fu, C. H. Y., & Gardner, M. (2021). Dehydration in older people: A systematic review of the effects of dehydration on health outcomes, healthcare costs and cognitive performance. Archives of gerontology and geriatrics, 95, 104380. https://doi.org/10.1016/j.archger.2021.104380
7. Garcia-Garcia D. (2022). Health Promotion and Hydration: A Systematic Review About Hydration Care. Florence Nightingale journal of nursing, 30(3), 310-321. https://doi.org/10.5152/FNJN.2022.21313.
8. Jimoh, F. O., Bunn, D., & Hooper, L. (2015). Assessment of a Self-Reported Drinks Diary for the Estimation of Drinks Intake by Care Home Residents: Fluid Intake Study in the Elderly (FISE). The journal of nutrition, health & aging, 19(5), 491-496. https://doi.org/10.1007/s12603-015-0458-3
9. Li, S., Xiao, X., & Zhang, X. (2023). Hydration Status in Older Adults: Current Knowledge and Future Challenges. Nutrients, 15(11), 2609. https://doi.org/10.3390/nu15112609
10. Lorenzo, I., Serra-Prat, M., & Yébenes, J. C. (2019). The Role of Water Homeostasis in Muscle Function and Frailty: A Review. Nutrients, 11(8), 1857. https://doi.org/10.3390/nu11081857.
11. Masot, O., Miranda, J., Santamaría, A. L., Paraiso Pueyo, E., Pascual, A., & Botigué, T.

(2020). Fluid Intake Recommendation Considering the Physiological Adaptations of Adults Over 65 Years: A Critical Review. Nutrients, 12(11), 3383. https://doi.org/10.3390/nu12113383 12. Mentes, J. C., & Gaspar, P. M. (2020). Hydration Management. Journal of gerontological nursing, 46(2), 19-30. https://doi.org/10.3928/00989134-20200108-03 13. Parkinson, E., Hooper, L., Fynn, J., Wilsher, S. H., Oladosu, T., Poland, F., Roberts, S., Van Hout, E., & Bunn, D. (2023). Low-intake dehydration prevalence in non-hospitalised older adults: Systematic review and meta-analysis. Clinical nutrition (Edinburgh,Scotland),42(8),1510-1520. https://doi.org/10.1016/j.clnu.2023.06.010 14. Paulis, S. J. C., Everink, I. H. J., Halfens, R. J. G., Lohrmann, C., & Schols, J. M. G. A. (2022). Dehydration in the nursing home: Recognition and interventions taken by Dutch nursing staff. Journal of advanced nursing, 78(4), 1044-1054. https://doi.org/10.1111/jan.15032 15. Purvis, S., & Gion, T. (2024). Fluid Status Vulnerability in Older Adults. Journal of infusion nursing: the official publication of the Infusion Nurses Society, 47(1), 49-53. https://doi.org/10.1097/NAN.0000000000000534 16. Siette, J., Berry, H., Jorgensen, M., Brett, L., Georgiou, A., McClean, T., … & Westbrook, J. (2020). Social participation among older adults receiving community care services. Journal of Applied Gerontology, 40(9), 997-1007. https://doi.org/10.1177/0733464820938973 17. Syed, S, Devlin, K, Andrade, A, Flanagan, K, Bruyn-Martin, L, Millar, V, Brown, S and Keller, H. (2024). Wet Your Whistle with Water (W3) to Improve Water Intake in Seniors' Care. Journal of Long-Term Care, , pp. 107-121. https://doi. org/10.31389/jltc.219 18. Veilleux, J. C., Caldwell, A. R., Johnson, E. C., Kavouras, S., McDermott, B. P., & Ganio, M. S. (2020). Examining the links between hydration knowledge, attitudes and behavior. European journal of nutrition, 59, 991-1000.

19. Volkert, D., Beck, A. M., Cederholm, T., Cruz-Jentoft, A., Goisser, S., Hooper, L., Kiesswetter, E., Maggio, M., Raynaud-Simon, A., Sieber, C. C., Sobotka, L., van Asselt, D., Wirth, R., & Bischoff, S. C. (2019). ESPEN guideline on clinical nutrition and hydration in geriatrics. Clinical nutrition (Edinburgh, Scotland), 38(1), 10-47. https://doi.org/10.1016/j.clnu.2018.05.024 20. Volkert D, Marie Beck A, Cederholm T, Cruz-Jentoft A, Hooper L, Kiesswetter E, Maggio M, Sieber C, Sobotka L, van Asselt D, Wirth R, Bischoff SC, Benoit F, De Breucker S, Raynaud-Simon A, Annweiler C, Sanchez-Rodriguez D. (2024). Guide pratique de la Société européenne de nutrition clinique : nutrition clinique et hydratation en gériatrie. Geriatr Psychol Neuropsychiatr Vieil; 22(3): 273-315. doi:10.1684/pnv.2024.1183

ELIGIBILITY:
Inclusion Criteria:

* Daily water and other fluid intake below the recommended levels: less than 2.0 L/day for older adult men and less than 1.6 L/day for older adult women (ESPEN Guidelines, 2024) Aged between 65 and 84 years Having at least a primary school education Having sufficient motor skills Having the cognitive capacity, willingness, and experience necessary to use technology Willing to participate in the study Owning a mobile phone compatible with the application Having prior experience using mobile applications

Exclusion Criteria:

* Diagnosed with moderate or severe cognitive impairment (MMSE < 24)
* Having vision or hearing impairments that prevent participation
* Diagnosed with advanced stage chronic kidney disease (Stage 4-5)
* Diagnosed with congestive heart failure (NYHA class III-IV)
* Being on fluid restriction by medical order
* Having a diagnosed urinary incontinence condition
* Having a diagnosis of terminal illness or active cancer treatment
* Participating in another hydration-related clinical study
* Experiencing a disruption in app usage for one week or longer for any reason

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Hydration Knowledge, Attitude, and Behavior Scale Scores | Baseline and 8 weeks after the intervention
  Participants' hydration-related knowledge, attitude, and behavior will be assessed using the Turkish version of the Hydration Knowledge, Attitude, and Behavior Scale (HyKS). The scale includes 16 knowledge items, 18 attitude items, and 4 behavior items. Scores are calculated separately for each domain. Higher scores indicate improved knowledge, more positive attitudes, and healthier hydration behaviors.

SECONDARY OUTCOMES:
System Usability Score of the Mobile Hydration Tracking Application | Week 4 and Week 8 after intervention
  Usability and user satisfaction with the hydration tracking mobile application will be assessed using the Turkish version of the System Usability Scale (SUS). The SUS consists of 10 items rated on a 5-point Likert scale. The total score is calculated by summing item scores after reverse scoring specific items (2, 4, 6, 8, and 10), then multiplying the result by 2.5 to yield a total score ranging from 0 to 100. Higher scores indicate better usability. Scores of 65-70 and above reflect acceptable usability. The SUS is a reliable, validated tool to assess user experience in mobile health interventions

OTHER OUTCOMES:
Fluid Intake Habits Based on Self-Reported Form | Baseline, Week 4, and Week 8
  Fluid intake habits will be assessed using a self-developed "Fluid Intake Habits Form" created by the investigator. The form collects descriptive data on the types and amounts of fluids consumed daily, frequency and timing of fluid intake, personal fluid intake goals, and behaviors such as self-monitoring. The form also identifies factors affecting fluid consumption (e.g., medication use, chronic illness, environmental influences). Expert opinion will obtained to validate the content. Responses will be analyzed to observe qualitative and quantitative changes in fluid intake patterns over the course of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Özlem KÜÇÜKGÜÇLÜ, Prof., Study Director — Dokuz Eylul University Faculty of Nursing

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) including scores from the Hydration Knowledge, Attitude, and Behavior Scale (HyKS), System Usability Scale (SUS), and self-reported fluid intake data will be shared with qualified researchers upon reasonable request.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: The IPD and supporting documentation will be available starting 6 months after publication of the main study results. Data will be accessible for a period of 5 years from that date.
Access Criteria: Access will be granted to qualified researchers affiliated with academic institutions or healthcare organizations, for the purpose of conducting meta-analyses or secondary analyses related to hydration behavior in older adults. Requests can be made by contacting the principal investigator via email. A data access agreement may be required.

REFERENCES:
- See also: Related Info — https://www.deu.edu.tr